CLINICAL TRIAL: NCT04521348
Title: A Phase II Study to Explore the Safety and Efficacy of Multiple Target Kinase Inhibitor(mTKI) Combined With Anti-Programmed Death-1(PD-1) Antibody in the Treatment of Advanced Thyroid Cancer
Brief Title: Multiple Target Kinase Inhibitor and Anti-Programmed Death-1 Antibody in Patients With Advanced Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ji Dongmei, Associated Professor, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ahead-T210
Record Dates: First submitted 2019-10-25; First posted 2020-08-20 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- RAIR-DTC arm (Experimental): Multiple Target Kinase Inhibitor(mTKI) Combined with Anti-Programmed Death-1(PD-1) Antibody
  Interventions: Drug: multiple tyrosine kinase inhibitor(mTKI) Combined with anti-PD-1 antibody
- MTC arm (Experimental): Multiple Target Kinase Inhibitor(mTKI) Combined with Anti-Programmed Death-1(PD-1) Antibody
  Interventions: Drug: multiple tyrosine kinase inhibitor(mTKI) Combined with anti-PD-1 antibody
- ATC arm (Experimental): Multiple Target Kinase Inhibitor(mTKI) Combined with Anti-Programmed Death-1(PD-1) Antibody
  Interventions: Drug: multiple tyrosine kinase inhibitor(mTKI) Combined with anti-PD-1 antibody
- DTC unsuitable for RAI arm (Experimental): Multiple Target Kinase Inhibitor(mTKI) Combined with Anti-Programmed Death-1(PD-1) Antibody
  Interventions: Drug: multiple tyrosine kinase inhibitor(mTKI) Combined with anti-PD-1 antibody

INTERVENTIONS:
Drug: multiple tyrosine kinase inhibitor(mTKI) Combined with anti-PD-1 antibody — Patients receive Multiple Target Kinase Inhibitor(mTKI) Combined with Anti-Programmed Death-1(PD-1) Antibody
  Other Names: mTKI, PD-1 antibody

SUMMARY:
The study is being conducted to evaluate the safety and efficacy of Multiple Target Kinase Inhibitor(mTKI) Combined with Anti-Programmed Death-1(PD-1) Antibody in subjects with advanced thyroid cancer.

DETAILED DESCRIPTION:
We will recruit four types of advanced thyroid cancer patients. Arm A will enroll the radioactive Iodine-refractory differentiated thyroid cancer(RAIR-DTC). Arm B will recruit the advanced medullary thyroid cancer(MTC). Arm C will include the advanced anaplastic thyroid cancer(ATC). Arm D will include the differentiated thyroid cancer that unsuitable for 131I treatment.

This clinical trial will be conducted under Simon's optimal two-stage design.

For arm A, the first stage needs 8 participants, if 4 or more participants acquire remission, the study will move on to the second stage and enroll another 16 patients to achieve a total number of 24 participants enrolled.

For arm B, the first stage needs 8 participants, if 4 or more participants acquire remission, the study will move on to the second stage and enroll another 16 patients to achieve a total number of 24 participants enrolled.

For arm C, the first stage needs 13 participants, if 4 or more participants acquire remission, the study will move on to the second stage and enroll another 30 patients to achieve a total number of 43 participants enrolled.

For arm D, the first stage needs 8 participants, if 4 or more participants acquire remission, the study will move on to the second stage and enroll another 16 patients to achieve a total number of 24 participants enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Patients volunteered to participate in this study and signed informed consent;
2. Age: ≥ 18 years old, male or female;
3. Advanced thyroid cancer patients couldn't be treated by local treatment such as surgery or microwave ablation, and are confirmed by histopathology or cytology to be one of the following three types of thyroid cancer:

   1. Local advanced or metastatic differentiated thyroid cancer, including papillary thyroid carcinoma (including follicular subtypes and poorly differentiated subtypes) and thyroid follicular carcinoma (including Hürthle cell subtypes, etc.).
   2. Local advanced or metastatic medullary thyroid carcinoma.
   3. Anaplastic thyroid cancer.
4. Differentiated thyroid cancer patients need to meet the definition of radioiodine refractory or is not suitable for 131I treatment. The definition of radioactive iodine refractory is as follows (meet one of the following conditions):

   1. At least one measurable lesion completely loses iodine uptake during radioiodine therapy;
   2. Although the lesion has iodine-receiving ability, at least one measurable lesion can still achieve progressive disease within 12 months after iodine131 treatment.
   3. has received a total dose of radioactive iodine therapy ≥ 22.2 GBq (≥ 600 mCi), and the final radioactive iodine therapy was within six months before enrollment;
5. If the subject is a patient with differentiated thyroid cancer, the TSH level should be at the inhibition level (<0.5 micro unit/L) from the screening period.
6. At least one measurable lesion (according to RECIST v1.1, long diameter of measurable lesion scanned by spiral CT should be ≥ 10 mm or short diameter of swollen lymph node should be ≥ 15 mm; according to RECIST vl.1 standards, a previously treated lesion with local treatment can be used as target lesions after clear progress);
7. Perfomance Status: 0~2;
8. Estimated survival time ≥ 12 weeks;
9. The main organs function are normal, and meet the following requirements (within 7 days before the start of study treatment):

   1. Blood routine examination(no blood transfusion within 14 days before screening, no granulocyte colony stimulating factor (G-CSF), no medication corrected):1) Hemoglobin (HB)≥ 90g / L;2) Neutrophil count (ANC) ≥ 1.5 × 109 / L;3) platelets (PLT) ≥ 80 × 109 / L;
   2. Blood biochemical tests are subject to the following criteria (no albumin is delivered 14 days prior to screening):1) Serum total bilirubin (BIL) ≤ 1.5 times the upper limit of normal (ULN); 2) alanine aminotransferase (ALT), aspartate aminotransferase (AST])< 2.5 × ULN; if liver metastasis, ALT and AST ≤ 5 × ULN;3) Serum creatinine (Cr) ≤ 1 × ULN or endogenous creatinine clearance > 50ml / min (Cockcroft-Gault formula);
   3. International normalized ratio (INR) ≤ 2.3 or prothrombin time (PT) exceeds the range of normal controls ≤ 6 seconds;
   4. Urine protein <2+ (if urine protein ≥ 2+, 24-hour urine protein can be quantified, 24-hour urine protein quantitation <1.0g can be included);
10. Women of childbearing age must have a negative pregnancy test (serum or urine) within 7 days prior to enrollment and volunteer to use appropriate methods during the observation period and within 8 weeks after the last study drug administration; for men, sterilization surgery should be performed, or agree to use appropriate methods of contraception during the observation period and within 8 weeks after the last administration of the study drug;
11. Patients voluntarily undergo tumor biopsy at the time of enrollment and out of the group.
12. Patient who are expected to have good compliance and can accept follow-up visit for the efficacy and adverse reactions according to the program requirements.

Exclusion Criteria:

1. Have other active malignancies within 5 years or at the same time. Localized tumors that have been cured, such as cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, superficial bladder cancer, prostate carcinoma in situ, cervical carcinoma in situ, and breast carcinoma in situ, can be enrolled.
2. Other anti-tumor treatments (including but not limited to chemotherapy, radiotherapy, etc.) were used within 28 days prior to the first use of the study drug. Except for thyroid stimulating hormone (TSH) inhibition therapy.
3. Patients who have previously been treated with immunological checkpoint inhibitors (including but not limited to Nivolumab, Pembrolizumab, Toripalimab, Sintilimab, etc.).
4. There are clinical symptoms or diseases of the heart that are not well controlled, such as:

   1. According to the New York Heart Association (NYHA) standard, level II or higher cardiac dysfunction or echocardiography: left ventricular ejection fraction<50%;
   2. unstable angina;
   3. Myocardial infarction occurred within 1 year before the start of treatment;
   4. Clinically significant supraventricular or ventricular arrhythmia that requires treatment or intervention;
   5. corrected QT interval(QTc) > 450ms (male); QTc > 470ms (female) (Calculation of QTc interval with Fridericia formula; if the QTc is abnormal, it can be detected three times at an interval of 2 minutes, and the average value is taken);
5. Patients with high blood pressure who cannot be reduced to normal range by antihypertensive medication (systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg) (average of BP based on ≥2 measurements), allowing the use of antihypertensive treatment to achieve the above parameters; there have been hypertensive crisis or hypertensive encephalopathy previously;
6. A variety of factors that affect the absorption of oral medications (such as inability to swallow, nausea and vomiting, chronic diarrhea and intestinal obstruction);
7. Patients with a risk of gastrointestinal bleeding may not be enrolled, including the following: (1) active digestive ulcer lesions, and fecal occult blood (++); (2) those with a history of melena and hematemesis within 3 months;
8. Abnormal coagulation function (INR>1.5×ULN,activated partial thromboplastin time>1.5×ULN), with bleeding tendency;
9. There is obvious hemoptysis within 2 months before screening, or hemoptysis volume is no less than half a teaspoon (2.5ml) per day;
10. Imaging studies have shown that the tumor has invaded important blood vessels or that the patient's tumor has a high probability of invading important blood vessels during treatment and causing fatal bleeding;
11. Thrombosis or embolic events occurred within 6 months prior to the start of treatment, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), pulmonary embolism, etc.
12. Currently associated with interstitial pneumonia or interstitial lung disease, or a history of interstitial pneumonia or interstitial lung disease requiring hormonal therapy, or other pulmonary fibrosis that may interfere with the assessment and management of immune-related pulmonary toxicity, Organized pneumonia (eg, bronchiolitis obliterans), pneumoconiosis, drug-associated pneumonia, idiopathic pneumonia, or evidence of active pneumonia or severe impaired lung function on a chest computed tomography (CT) scan during screening, but radiation pneumonitis is allowed in field of radiation: active tuberculosis;
13. There is autoimmune disease or a history of active autoimmune disease which may recur (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, pituitary inflammation, vasculitis, nephritis); patients who have skin diseases that do not require systemic treatment such as vitiligo, psoriasis, hair loss, patients who have controlled type 1 diabetes by using insulin, and patients who have completely relieved asthma in childhood and needn't intervention after be adults can be included; Asthmatic patients need bronchodilators for medical intervention cannot be included;
14. Use immunosuppressive agents or systemic hormonal therapy for immunosuppression within 14 days prior to initiation of study treatment (dose > 10 mg/day of prednisone or other therapeutic hormones);
15. Use strong CYP3A4/CYP2C19 inducers including rifampicin (and its analogs) and hyperforin perforatum or strong CYP3A4/CYP2C19 inhibitors within 14 days prior to initiation of study treatment;
16. Have a severe allergic history of any monoclonal antibody, anti-angiogenic targeted drug;
17. Uncontrolled infections during screening;
18. Pregnant or lactating women;
19. Patients refused to undergo a biopsy of the tumor at the time of enrollment and out of the group.
20. Other patients evaluated by physician to be unfit for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | Up to approximately 12 weeks
  Complete remission rate+ partial remission rate

SECONDARY OUTCOMES:
Duration of Response(DOR) | up to approximately 3 years
  Time from the date of first partial remission or complete remission to the date of disease progression, or death of any cause, or date of lost follow-up, whichever comes first, otherwise subject data were censored at time last known disease free.
Disease Control Rate(DCR) | Up to approximately 12 weeks
  Complete remission rate+ partial remission rate+stable disease rate
Time to response(TTR) | up to approximately 12 weeks
  Time from the initiation of the treatment to the first remission
Progression Free Survival(PFS) | up to approximately 3 years
  Time from the date of enrollment to of disease progression, or death of any cause, or date of lost follow-up, whichever comes first, otherwise subject data were censored at time last known disease free.
Overall survival(OS) | up to approximately 3 years
  Time from the date of enrollment to data of death from any cause, or date of lost follow-up, whichever comes first, and otherwise censored at time last known alive.
6-month overall survival rate | From the start of treatment to 6 months
  proportion of patients who lived 6 months or more since enrollment
12-month overall survival rate | From the start of treatment to 12 months
  proportion of patients who lived 12 months or more since enrollment
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | from the first drug administration to within 90 days for the last Anti-Programmed Death-1 Antibody dose
  incidence of treatment-related AEs and grade3/4 AEs according to CTCAE v4.0
Rate of dose suspension, dose reduction and dose termination | up to approximately 2 years
  proportion of patients who have experienced dose suspension, dose reduction and dose termination
Rate of dose reduction | up to approximately 2 years
  proportion of patients who have experienced dose reduction
Rate of dose termination | up to approximately 2 years
  proportion of patients who have experienced dose termination

CONTACTS AND LOCATIONS:
Overall Officials: JI DONGMEI, M.D, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China